CLINICAL TRIAL: NCT00577343
Title: Hospital Acquired and Community Acquired Methicillin Resistant Staph Aureus in the Outpatient Gastrointestinal Lab: A Prospective Study of Prevalence
Brief Title: Hospital Acquired and Community Acquired MRSA in GI Lab
Status: Withdrawn | Type: Observational
Why Stopped: study lacked funding to recruit
Sponsor: Indiana University (Other)
Responsible Party: Dr. Julia LeBlanc, Indiana University
Other Study IDs: 0705-31
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Hospital Acquired MRSA; Community Acquired MRSA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — buccal swab for saliva
Oversight: Data Monitoring Committee: No

SUMMARY:
Hospital acquired and community acquired methicillin resistant staph aureus (MRSA) has become an important health issue for in recent years. Up to two thirds of patients that are hospitalized may be colonized with MRSA. The prevalence in the community is also on the rise and affects the young and healthy. It is unclear what the true prevalence of MRSA is in our own hospital and outpatient setting. This information would be relevant to how healthcare staff adhere to contact and universal precautions. : The purpose of this study is to determine the prevalence of MRSA in patients that have gastrointestinal endoscopy and endoscopic ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* No evidence of dementia or altered mental status that would prohibit the giving and understanding of informed consent, and no evidence of psychiatric risk that would preclude adequate compliance with this protocol.

Subjects must provide signed written informed consent.

Exclusion Criteria:

* Inability to provide written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: gastrointestinal lab of oupatient and inpatients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The objective of this prospective study is to identify the prevalence of MRSA in patients that use the Indiana University GI lab. | less than one year

CONTACTS AND LOCATIONS:
Locations (1):
- Clarian/Indiana University Hospital, Indianapolis, Indiana, United States